CLINICAL TRIAL: NCT01827371
Title: A Phase II, Randomized, Open-Label Study to Evaluate the Safety and Immunogenicity of IMVAMUNE® Using Three Immunization Schedules and Two Modes of Delivery
Brief Title: Phase II Trial to Assess Safety and Immunogenicity of IMVAMUNE®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-0021; HHSN272200800004C
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2015-05

CONDITIONS: Smallpox
Keywords: Smallpox, vaccine, IMVAMUNE, Stratis, parent protocol
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

ARMS (4):
- Arm C (Experimental): 88 subjects receive IMVAMUNE® 1x10^8 TCID50/0.5 mL subcutaneously (SC) via syringe and needle on Days 1 and 22.
  Interventions: Biological: MVA Smallpox Vaccine
- Arm B (Experimental): 88 subjects receive IMVAMUNE® 1x10^8 TCID50/0.5 mL subcutaneously (SC) via syringe and needle on Days 1 and 15.
  Interventions: Biological: MVA Smallpox Vaccine
- Arm A (Experimental): 88 subjects receive IMVAMUNE® 1x10^8 TCID50/0.5 mL subcutaneously (SC) via syringe and needle on Days 1 and 29.
  Interventions: Biological: MVA Smallpox Vaccine
- Arm D (Experimental): 88 subjects receive IMVAMUNE® 1x10^8 TCID50/0.5 mL subcutaneously (SC) via Stratis™ on Days 1 and 29.
  Interventions: Biological: MVA Smallpox Vaccine

INTERVENTIONS:
Biological: MVA Smallpox Vaccine — Subjects receive two dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL per dose) via the SC route using either a syringe and needle or the Stratis™ system. Arm A receives doses via syringe and needle on days 1 and 29; Arm B receives doses via syringe and needle on days 1 and 15, Arm C receives doses via syringe and needle on days 1 and 22, Arm D receives doses via Stratis on days 1 and 29.

SUMMARY:
Imvamune (licensed name of MVA being developed as a smallpox vaccine) has been tested in over 2,000 individuals and is on path for licensure. This study will be a Phase II to evaluate three different immunization schedules and two different modes of delivery. The study will look at condensed schedules. Study will randomize subjects to one of four arms.

DETAILED DESCRIPTION:
This is a Phase II, randomized, open-label immunogenicity and safety study of different immunization schedules and delivery systems (syringe and needle vs. the Stratis™) in healthy, vaccinia-naïve adults 18 years to 40 years of age, inclusive. Approximately 352 subjects will be enrolled and randomized to one of four study arms. Study Arm A (N=88) will receive a two dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL per dose) via the SC route using a syringe and needle on Day 1 and 29. Study Arm B (N=88) will receive a two dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL per dose) via the SC route using a syringe and needle on Day 1 and 15. Study Arm C (N=88) will receive a two dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL) via the SC route using a syringe and needle on Day 1 and 22. Study Arm D (N=88) will receive a two dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL) via the SC route using the Stratis™ on Day 1 and 29. Immunogenicity assessments will be performed using ELISA and PRNT. Safety assessments will be done via solicited injection site and systemic reactions. Unsolicited AEs will be collected until 28 days post last injection and SAEs for the duration of the subjects' study participation. Safety laboratory assessments will be performed at baseline and 14 days after each vaccination. Primary outcome measures: For each subject, the peak PRNT will be defined as the highest titer among all available measurements post second vaccination; Occurrence of solicited local injection site reactions in subjects receiving vaccine via the Stratis™ compared to syringe and needle administration as collected on the memory aid and by in clinic assessment. Parent protocol to sub-study 13-0027.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 40 years of age, inclusive.
2. Read, signed, and dated informed consent document.
3. Available for follow-up for the planned duration of the study (six months after last immunization).
4. Acceptable medical history by screening evaluation and limited physical assessment.
5. If the subject is female and of childbearing potential, negative serum or urine pregnancy test at screening and within 24 hours prior to vaccination.
6. If the subject is female and of childbearing potential*, she agrees to practice abstinence** or use acceptable contraception*** through 56 days after the last vaccination in order to avoid pregnancy:

   * a woman is considered of childbearing potential unless post-menopausal (>/= 1 year without menses) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy)

   **No sexual intercourse with men (vaginal penetration by a penis, coitus)

   ***Acceptable contraception methods are restricted to effective devices (IUDs, NuvaRing®) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, condoms with spermicidal agents, monogamous relationship with a vasectomized partner who has been vasectomized for 6 months or more prior to study entry, or successful Essure placement with documented confirmation test at least 3 months after the procedure, and any other FDA-approved contraceptive method
7. Negative test for HIV.
8. Alanine Aminotransferase (ALT) <1.25 times the central lab upper limit of normal.
9. Negative hepatitis B surface antigen and negative antibody to hepatitis C virus.
10. Negative urine glucose and negative or trace urine protein by dipstick or urinalysis.
11. Adequate renal function (defined as a serum creatinine not exceeding the central lab's upper limit of normal).
12. Electrocardiogram (ECG) with no clinically significant abnormalities*

    * e.g., complete left or right bundle branch block, incomplete left bundle branch block or sustained ventricular arrhythmia, or two PVC's in a row, or ST elevation consistent with ischemia)
13. Acceptable hematology parameters:

    * Hemoglobin (Hgb) equal or above the lower limit of central lab normal (sex-specific);
    * White Blood Cell (WBC) > 3,800 and < 10,900/mm^3;
    * Platelets >/=120,000/mm^3
14. Body mass index >/=18.5-< 35.
15. Be able to understand and comply with planned study procedures.

Exclusion Criteria:

1. History of immunodeficiency.
2. Typical vaccinia scar.
3. Known or suspected history of smallpox vaccination including MVA alone or as a vector, as well as other investigational smallpox vaccines.
4. Military service prior to 1991 or after January 2003.
5. Known or suspected significant underlying illness including, but not limited to, clinically significant liver disease, diabetes mellitus, or moderate to severe kidney impairment.
6. Malignancy (not including squamous cell skin cancer or basal cell skin cancer unless at the vaccination site) or history of skin cancer at the vaccination site.
7. Active autoimmune disease. Persons with vitiligo or thyroid disease (e.g., taking thyroid hormone replacement) are not excluded.
8. History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor*

   *Subjects with a not clinically relevant heart murmur, i.e., without any pathological ECG/arrhythmias or under treatment are not excluded.
9. Systolic blood pressure >/= 150mmHg or diastolic blood pressure >/= 100mmHg.
10. Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's (NCEP) risk assessment tool*

    *NOTE that this criterion applies only to subjects 20 years of age and older AND only if at least one of the following apply:
    * have smoked a cigarette in the past month, and/or
    * have hypertension (defined as systolic blood pressure >140 mm Hg) or are on antihypertensive medication, and/or
    * have a family history of coronary heart disease in male first-degree relative (father or brother) <55 years of age or a female first-degree relative (mother or sister) <65 years of age

    URL for NCEP risk assessment tool: http://cvdrisk.nhlbi.nih.gov/calculator.asp (if a subject has an HDL of greater than 100mg/dl please enter 100 in the tool)
11. High-dose corticosteroid use for greater than 2 weeks duration within three months prior to vaccination or current use of immunosuppressive medication:

    * >5 mg prednisone or equivalent is considered high dose and immunosuppressive
    * Corticosteroid nasal sprays for allergic rhinitis are permissible
    * Persons who are using a topical steroid for mild uncomplicated dermatitis such as poison ivy or contact dermatitis may be enrolled the day after their therapy is completed
    * Inhaled steroids for asthma are not permissible
    * Oral/parenteral corticosteroids given for non-chronic conditions not expected to recur are permissible if the length of therapy was </= 14 days with completion at least 30 days prior to enrollment.
12. Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol.
13. Any history of illegal injection drug use.
14. Receipt or planned receipt of inactivated vaccine from 14 days prior to the first vaccination through 14 days post second vaccination.
15. Receipt or planned receipt of any other live attenuated vaccine within 30 days prior to the first vaccination through 30 days post second vaccination.
16. Use of any other experimental agent within 30 days prior to vaccination and for the duration of the subject's participation in the study.
17. Receipt of blood products or immunoglobulin, including Rhogam, within six months prior to vaccination.
18. Donation of a unit of blood within 56 days prior to vaccination or planned donation prior to 28-days following the last vaccination.
19. Pregnant or breastfeeding women.
20. Active exfoliative skin disorders/conditions, current varicella zoster virus infection, or any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2×2 cm.
21. Any condition that, in the opinion of the investigator, might interfere with assessing the study objectives.
22. Known allergy to egg, aminoglycoside (including gentamicin) or chicken.
23. Study personnel.
24. Allergic reaction to any vaccine.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 435 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - University of Maryland Medical System - General Clinical Research Center (GCRC), Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle - Vaccines and Infectious Diseases, Seattle, Washington

REFERENCES:
- [Derived] Jackson LA, Frey SE, El Sahly HM, Mulligan MJ, Winokur PL, Kotloff KL, Campbell JD, Atmar RL, Graham I, Anderson EJ, Anderson EL, Patel SM, Fields C, Keitel W, Rouphael N, Hill H, Goll JB. Safety and immunogenicity of a modified vaccinia Ankara vaccine using three immunization schedules and two modes of delivery: A randomized clinical non-inferiority trial. Vaccine. 2017 Mar 23;35(13):1675-1682. doi: 10.1016/j.vaccine.2017.02.032. Epub 2017 Feb 27. PMID 28256358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult males and females recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 17JUN2013 and 23SEP2014.
Groups:
- Arm A: IMVAMUNE Days 1+29, Syringe and Needle: IMVAMUNE 1x10^8 TCID50/0.5 mL subcutaneously (SC) via syringe and needle on Days 1 and 29.
- Arm B: IMVAMUNE Days 1+15, Syringe and Needle: IMVAMUNE 1x10^8 TCID50/0.5 mL SC) via syringe and needle on Days 1 and 15.
- Arm C: IMVAMUNE Days 1+22, Syringe and Needle: IMVAMUNE 1x10^8 TCID50/0.5 mL subcutaneously (SC) via syringe and needle on Days 1 and 22.
- Arm D: IMVAMUNE Days 1+29, Stratis: IMVAMUNE® 1x10^8 TCID50/0.5 mL subcutaneously (SC) via Stratis™ auto injector on Days 1 and 29.
Period: Overall Study
Arm/Group | Arm A: IMVAMUNE Days 1+29, Syringe and Needle | Arm B: IMVAMUNE Days 1+15, Syringe and Needle | Arm C: IMVAMUNE Days 1+22, Syringe and Needle | Arm D: IMVAMUNE Days 1+29, Stratis
Started | 115 | 96 | 104 | 120
Completed | 102 | 89 | 93 | 97
Not Completed | 13 | 7 | 11 | 23
Not completed — Adverse Event | 0 | 0 | 4 | 2
Not completed — Lost to Follow-up | 0 | 2 | 0 | 4
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 1
Not completed — Temporary study halt to vaccinations | 11 | 2 | 5 | 13

BASELINE CHARACTERISTICS:
Population: All participants are included in the baseline analysis population
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: IMVAMUNE Days 1+29, Syringe and Needle | Arm B: IMVAMUNE Days 1+15, Syringe and Needle | Arm C: IMVAMUNE Days 1+22, Syringe and Needle | Arm D: IMVAMUNE Days 1+29, Stratis | Total
Number analyzed (Participants) | 115 | 96 | 104 | 120 | 435
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 115 | 96 | 104 | 120 | 435
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (5.6) | 27.1 (5.4) | 27.2 (5.0) | 27.9 (5.2) | 27.4 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 49 | 59 | 60 | 229
  Male | 54 | 47 | 45 | 60 | 206
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 12 | 7 | 33
  Not Hispanic or Latino | 104 | 92 | 92 | 113 | 401
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 3 | 7 | 12 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 20 | 15 | 17 | 18 | 70
  White | 81 | 70 | 74 | 86 | 311
  More than one race | 6 | 8 | 4 | 4 | 22
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 115 | 96 | 104 | 120 | 435

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Peak Plaque Reduction Neutralization Titer (PRNT) After Second Vaccination
Description: Blood was collected from all participants at 8, 15, 22 and 29 days after receipt of the second vaccination for assessment of plaque reduction neutralization titers. The peak titer for each participant was defined as the highest titer among all available measurements post second vaccination. The geometric mean for each group was then assessed from individual participants' peak titers.
Time Frame: Day 7 through Day 31 after 2nd vaccination
Population: The modified ATP population was defined as all participants who received both vaccinations in window, excluding those who did not have a complete dose delivered or received non-study vaccinations. Only measurements (blood draws) between Days 7-31 were considered and subjects had to have at least two measurements in that range to be included.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Arm A: IMVAMUNE Days 1+29, Syringe and Needle | Arm B: IMVAMUNE Days 1+15, Syringe and Needle | Arm C: IMVAMUNE Days 1+22, Syringe and Needle | Arm D: IMVAMUNE Days 1+29, Stratis
Number analyzed (Participants) | 84 | 85 | 84 | 79
titers | 138.0 [110.1 to 172.8] | 55.1 [42.3 to 71.7] | 75.9 [58.5 to 98.4] | 103.5 [80.8 to 132.6]
Statistical Analysis 1: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm B: IMVAMUNE Days 1+15, Syringe and Needle; Hypotheses: H0: log2(GMT(Arm A))-log2 (GMT(Arm B)) ≥ 1 or GMT(Arm A)/GMT (Arm B) ≥2 H1: log2(GMT(Arm A))-log2(GMT(Arm B)) < 1 or GMT(Arm A)/GMT(Arm B) < 2. Sample Size: The SD for log2 PRNT based on a prior study was~1.9. The margin of non-inferiority was specified as a 2-fold difference on the original scale (1 on the log2 scale). The objective included three non-inferiority evaluations (A vs. B, A vs. C, A vs. D). Thus, a Bonferroni-corrected alpha of 2.5% / 3 = 0.833% was used. Power=80%; Test type: Non-Inferiority or Equivalence — Hypotheses Evaluation: The difference between the mean log2 peak titer for the control arm (Study Arm A) and each investigational arm (Study Arm B, C, or D) and the associated two sided 98.33% confidence intervals (CI) for the estimated population mean difference were calculated. If the upper limit of the 98.33% CI was less than 1, Study Arm B, C or D was considered to be non-inferior to Study Arm A; Mean Difference (Log2 Scale) = 1.32, 98.33% CI 2-sided [0.72 to 1.93]
Statistical Analysis 2: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm C: IMVAMUNE Days 1+22, Syringe and Needle; Hypotheses: H0: log2(GMT(Arm A))-log2 (GMT(Arm C)) ≥ 1 or GMT(Arm A)/GMT (Arm C) ≥2 H1: log2(GMT(Arm A))-log2(GMT(Arm C)) < 1 or GMT(Arm A)/GMT(Arm C) < 2. Sample Size: The SD for log2 PRNT based on a prior study was~1.9. The margin of non-inferiority was specified as a 2-fold difference on the original scale (1 on the log2 scale). The objective included three non-inferiority evaluations (A vs. B, A vs. C, A vs. D). Thus, a Bonferroni-corrected alpha of 2.5% / 3 = 0.833% was used. Power=80%; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Log2 Scale) = 0.86, 98.33% CI 2-sided [0.26 to 1.47]
Statistical Analysis 3: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm D: IMVAMUNE Days 1+29, Stratis; Hypotheses: H0: log2(GMT(Arm A))-log2 (GMT(Arm D)) ≥ 1 or GMT(Arm A)/GMT (Arm D) ≥2 H1: log2(GMT(Arm A))-log2(GMT(Arm D)) < 1 or GMT(Arm A)/GMT(Arm D) < 2. Sample Size: The SD for log2 PRNT based on a prior study was~1.9. The margin of non-inferiority was specified as a 2-fold difference on the original scale (1 on the log2 scale). The objective included three non-inferiority evaluations (A vs. B, A vs. C, A vs. D). Thus, a Bonferroni-corrected alpha of 2.5% / 3 = 0.833% was used. Power=80%; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Log2 Scale) = 0.41, 98.33% CI 2-sided [-0.17 to 1.0007]

2. Primary Outcome: Percentage of Participants Reporting Moderate or Severe Solicited Local Injection Site Reactions After Receiving Vaccine Via the Stratis™ Compared to Syringe and Needle Administration
Description: Participants maintained a memory aid to record daily the occurrence of local injection site reactions for 15 days after vaccination based on their interference with daily activities (pain and itchiness at injection site, underarm pain and swelling) or based on a quantitative measurement of the reaction (redness, swelling). In the subjective grading scale, severe reactions prevented daily activities, moderate reactions interfered with but did not prevent daily activities, and mild reactions were present but did not interfere with daily activities. For the quantitative scale, severe reactions greater than 30 millimeters (mm), moderate reactions were 15-30mm, and mild reactions were 1-15mm. Participants are counted by the maximum severity on any of the 15 days, and for this outcome measure, only those reporting moderate or severe events are counted. Formal comparisons by Fisher's Exact test were conducted for Arm D (Stratis, Day 1,29) compared to A
Time Frame: 15 days after each vaccination
Population: All subjects receiving at least one vaccination are included in the analysis population 'as treated', so one subject randomized to Arm C vaccinated out of window, equivalent to the schedule for Arm A, was analyzed for this outcome measure as Arm A.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: IMVAMUNE Days 1+29, Syringe and Needle | Arm B: IMVAMUNE Days 1+15, Syringe and Needle | Arm C: IMVAMUNE Days 1+22, Syringe and Needle | Arm D: IMVAMUNE Days 1+29, Stratis
Number analyzed (Participants) | 116 | 96 | 103 | 120
percentage of participants
  Pain at Injection Site | 28 | 36 | 26 | 33
  Itchiness at Injection Site | 6 | 10 | 17 | 12
  Underarm Pain | 4 | 4 | 3 | 5
  Underarm Swelling | 2 | 2 | 2 | 1
  Redness at Injection Site | 54 | 52 | 60 | 79
  Swelling at Injection Site | 52 | 47 | 52 | 70
  Any Solicited Local Symptom | 73 | 69 | 77 | 90
Statistical Analysis 1: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm D: IMVAMUNE Days 1+29, Stratis; Hypothesis: H0: Pr('Pain at Injection Site ' Arm A) = Pr('Pain at Injection Site ' Arm D) H1: Pr('Pain at Injection Site ' Arm A) not = Pr('Pain at Injection Site ' Arm D); Test type: Superiority or Other; p = 0.4782, Fisher Exact — alpha= 5%
Statistical Analysis 2: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm D: IMVAMUNE Days 1+29, Stratis; Hypothesis: H0: Pr('Itchiness at Injection Site' Arm A) = Pr('Itchiness at Injection Site' Arm D) H1: Pr('Itchiness at Injection Site' Arm A) not = Pr('Itchiness at Injection Site' Arm D); Test type: Superiority or Other; p = 0.1704, Fisher Exact — alpha= 5%
Statistical Analysis 3: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm D: IMVAMUNE Days 1+29, Stratis; Hypothesis: H0: Pr('Underarm pain' Arm A) = Pr('Underarm pain' Arm D) H1: Pr('Underarm pain' Arm A) not = Pr('Underarm pain' Arm D); Test type: Superiority or Other; p = 1.000, Fisher Exact — alpha= 5%
Statistical Analysis 4: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm D: IMVAMUNE Days 1+29, Stratis; Hypothesis: H0: Pr('Underarm swelling' Arm A) = Pr('Underarm swelling' Arm D) H1: Pr('Underarm swelling' Arm A) not = Pr('Underarm swelling' Arm D); Test type: Superiority or Other; p = 0.6171, Fisher Exact — alpha= 5%
Statistical Analysis 5: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm D: IMVAMUNE Days 1+29, Stratis; Hypothesis: H0: Pr('Redness at Injection Site' Arm A) = Pr('Redness at Injection Site' Arm D) H1: Pr('Redness at Injection Site' Arm A) not = Pr('Redness at Injection Site' Arm D); Test type: Superiority or Other; p < 0.0001, Fisher Exact — alpha=5%
Statistical Analysis 6: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm D: IMVAMUNE Days 1+29, Stratis; Hypothesis: H0: Pr('Swelling at Injection Site' Arm A) = Pr('Swelling at Injection Site' Arm D) H1: Pr('Swelling at Injection Site' Arm A) not = Pr('Swelling at Injection Site' Arm D); Test type: Superiority or Other; p = 0.0050, Fisher Exact — alpha=5%
Statistical Analysis 7: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm D: IMVAMUNE Days 1+29, Stratis; Hypothesis: H0: Pr('Any Solicited Local Reaction' Arm A) = Pr('Any Solicited Local Reaction' Arm D) H1: Pr('Any Solicited Local Reaction' Arm A) not = Pr('Any Solicited Local Reaction' Arm D); Test type: Superiority or Other; p = 0.0012, Fisher Exact — alpha=5%

3. Secondary Outcome: Geometric Mean Peak ELISA Titer After Second Vaccination
Description: Blood was collected from all participants at 8, 15, 22 and 29 days after receipt of the second vaccination for assessment of antibody titers by ELISA. The peak titer for each participant was defined as the highest titer among all available measurements post second vaccination. The geometric mean for each group was then assessed from individual participants' peak titers.
Time Frame: Day 7 through 31 after the 2nd vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Arm A: IMVAMUNE Days 1+29, Syringe and Needle | Arm B: IMVAMUNE Days 1+15, Syringe and Needle | Arm C: IMVAMUNE Days 1+22, Syringe and Needle | Arm D: IMVAMUNE Days 1+29, Stratis
Number analyzed (Participants) | 84 | 85 | 84 | 79
titers | 1259.8 [1093.0 to 1451.9] | 741.4 [625.0 to 879.6] | 1021.0 [878.1 to 1187.1] | 1351.8 [1130.0 to 1617.1]
Statistical Analysis 1: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm B: IMVAMUNE Days 1+15, Syringe and Needle; Hypotheses: H0: log2(GMT(Arm A))-log2 (GMT(Arm B)) ≥ 1 or GMT(Arm A)/GMT (Arm B) ≥2 H1: log2(GMT(Arm A))-log2(GMT(Arm B)) < 1 or GMT(Arm A)/GMT(Arm B) < 2. The margin of non-inferiority was specified as a 2-fold difference on the original scale (1 on the log2 scale). The objective included three non-inferiority evaluations (A vs. B, A vs. C, A vs. D). Thus, a Bonferroni-corrected alpha of 2.5% / 3 = 0.833% was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Log2 Scale) = 0.76, 98.33% CI 2-sided [0.37 to 1.15]
Statistical Analysis 2: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm C: IMVAMUNE Days 1+22, Syringe and Needle; Hypotheses: H0: log2(GMT(Arm A))-log2 (GMT(Arm C)) ≥ 1 or GMT(Arm A)/GMT (Arm C) ≥2 H1: log2(GMT(Arm A))-log2(GMT(Arm C)) < 1 or GMT(Arm A)/GMT(Arm C) < 2. The margin of non-inferiority was specified as a 2-fold difference on the original scale (1 on the log2 scale). The objective included three non-inferiority evaluations (A vs. B, A vs. C, A vs. D). Thus, a Bonferroni-corrected alpha of 2.5% / 3 = 0.833% was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Log2 Scale) = 0.30, 98.33% CI 2-sided [-0.06 to 0.67]
Statistical Analysis 3: Comparison: Arm A: IMVAMUNE Days 1+29, Syringe and Needle vs Arm D: IMVAMUNE Days 1+29, Stratis; Hypotheses: H0: log2(GMT(Arm A))-log2 (GMT(Arm D)) ≥ 1 or GMT(Arm A)/GMT (Arm D) ≥2 H1: log2(GMT(Arm A))-log2(GMT(Arm D)) < 1 or GMT(Arm A)/GMT(Arm D) < 2. The margin of non-inferiority was specified as a 2-fold difference on the original scale (1 on the log2 scale). The objective included three non-inferiority evaluations (A vs. B, A vs. C, A vs. D). Thus, a Bonferroni-corrected alpha of 2.5% / 3 = 0.833% was used; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mean Difference (Log2 Scale) = -0.10, 98.33% CI 2-sided [-0.50 to 0.30]

4. Secondary Outcome: Number of Subjects Experiencing Serious Adverse Events (SAEs) Associated With IMVAMUNE
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation thereof; was a congenital anomaly/birth defect; or may have jeopardized the participant, or required intervention to prevent one of the outcomes. Association with IMVAMUNE was determined by the investigator and defined as "Related", meaning a reasonable possibility that the study product caused the adverse event. Reasonable possibility was defined as there being evidence to suggest a causal relationship between the study product and the adverse event.
Time Frame: Day 1 after the first vaccination through 180 days after the 2nd vaccination.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Arm A: IMVAMUNE Days 1+29, Syringe and Needle | Arm B: IMVAMUNE Days 1+15, Syringe and Needle | Arm C: IMVAMUNE Days 1+22, Syringe and Needle | Arm D: IMVAMUNE Days 1+29, Stratis
Number analyzed (Participants) | 116 | 96 | 103 | 120
participants | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 15 days after each vaccination, unsolicited non-serious AEs through 28 days after last vaccination, and SAEs through 180 days after last vaccination.
Description: Subjects were analyzed as treated for the safety population, so one subject randomized to Arm C but vaccinated out of window, equivalent to the schedule for Arm A, was analyzed as an Arm A subject.
Arm/Group | Arm A: IMVAMUNE Days 1+29, Syringe and Needle | Arm B: IMVAMUNE Days 1+15, Syringe and Needle | Arm C: IMVAMUNE Days 1+22, Syringe and Needle | Arm D: IMVAMUNE Days 1+29, Stratis
Serious Adverse Events (participants affected / at risk) | 2/116 | 1/96 | 1/103 | 1/120
Other Adverse Events (participants affected / at risk) | 114/116 | 94/96 | 103/103 | 119/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: IMVAMUNE Days 1+29, Syringe and Needle (N=116) | Arm B: IMVAMUNE Days 1+15, Syringe and Needle (N=96) | Arm C: IMVAMUNE Days 1+22, Syringe and Needle (N=103) | Arm D: IMVAMUNE Days 1+29, Stratis (N=120)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type I hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: IMVAMUNE Days 1+29, Syringe and Needle (N=116) | Arm B: IMVAMUNE Days 1+15, Syringe and Needle (N=96) | Arm C: IMVAMUNE Days 1+22, Syringe and Needle (N=103) | Arm D: IMVAMUNE Days 1+29, Stratis (N=120)
HEADACHE (Nervous system disorders) | 12 (12) | 6 (8) | 13 (16) | 15 (17)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 (10) | 5 (6) | 11 (11) | 11 (11)
VACCINATION SITE BRUISING (General disorders) | 4 (4) | 1 (1) | 4 (4) | 9 (9)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 18 (19) | 20 (25) | 17 (23) | 21 (27) — Solicited on the subject memory aid as "Joint pain"
APPETITE DISORDER (Metabolism and nutrition disorders) | 19 (21) | 16 (18) | 14 (14) | 19 (21) — Solicited on the subject memory aid as 'Change in appetite'
CHILLS (General disorders) | 10 (11) | 16 (19) | 13 (16) | 21 (23)
MALAISE (General disorders) | 56 (76) | 59 (84) | 49 (65) | 61 (79) — Solicited on the memory aid as "Feeling tired"
MYALGIA (Musculoskeletal and connective tissue disorders) | 42 (59) | 49 (66) | 46 (57) | 49 (63) — Solicited on the memory aid as "Muscle aches"
NAUSEA (Gastrointestinal disorders) | 20 (23) | 15 (17) | 19 (22) | 20 (21)
INJECTION SITE OEDEMA (General disorders) | 74 (111) | 67 (107) | 74 (114) | 112 (183) — Solicited on the memory aid as "Edema/swelling measurement", reported as experienced if size >0mm
INJECTION SITE ERYTHEMA (General disorders) | 82 (124) | 66 (109) | 81 (126) | 114 (185) — Solicited on the memory aid as "Erythema/redness measurement", reported as experienced if size >0mm
INJECTION SITE PRURITUS (General disorders) | 67 (87) | 44 (64) | 52 (76) | 86 (124) — Solicited on the memory aid as "Itchiness at injection site"
INJECTION SITE PAIN (General disorders) | 108 (173) | 84 (153) | 96 (154) | 115 (183) — Solicited by memory aid as "Pain at injection site"
AXILLARY PAIN (General disorders) | 17 (20) | 21 (30) | 18 (20) | 28 (35) — Solicited on the memory aid as "Underarm pain"
LOCAL SWELLING (General disorders) | 11 (11) | 14 (19) | 16 (18) | 19 (20) — Solicited on the memory aid as "Underarm swelling"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less